CLINICAL TRIAL: NCT05290909
Title: The Effectiveness of Blended and Problem-based Learning to Improve the Geriatric Nursing of Critical Thinking and Ethical Competence Among Nursing Students
Brief Title: The Effectiveness of Blended and Problem-based Learning to Improve the Competence of Geriatric Nursing Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Chia Jung Hsieh, Ph.D., RN, Associate Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FJU-IRB C110071
Record Dates: First submitted 2022-03-12; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Narrative Ethics
Keywords: Nursing students; blended model; problem-based learning; critical thinking; ethical competence
MeSH Terms: conditions — Narration | interventions — WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The protocol of blended and problem-based learning (Experimental): The experimental group will accept the protocol of blended and problem-based learning in the professional ethics course, 2 hours /per week, for 18 weeks
  Interventions: Other: The protocol of blended and problem-based learning
- The traditional problem-oriented teaching model (Active Comparator): The control group will accept the traditional problem-oriented teaching model in the professional ethics course, 2 hours /per week, for 18 weeks
  Interventions: Other: The traditional problem-oriented teaching model

INTERVENTIONS:
Other: The protocol of blended and problem-based learning — The protocol of blended and problem-based learnin: The online platforms used in this research are the school's iLMS platform, online digital learning, and online opinion exchange platform. It will use online resources (Google, open educational resources, YouTube copyrighted medical micro-movies, and audio-visual materials), and the theme will be elderly care or emerging Multimedia resources on infectious themes, as well as real-time interaction with kahoot or Slido electronic whiteboards, will be uploaded to the office3655The One website. Drive is provided by the school (the school account is used to store course resources) and the system of digital theoretical course concepts in advance. Broadcasting, video (such as: values and conflicts; ethics and morality; patient rights and responsibilities; nurses' rights and responsibilities; ethical theory; basic ethical principles; ethical dilemmas and ethical decision-making; etc.), pre-recorded and stored on the Internet Road platform iLMS.
  Other Names: The experimental group will accept the protocol of blended and problem-based learning in the professional ethics course, 2 hours /per week, for 18 weeks
  Arms: The protocol of blended and problem-based learning
Other: The traditional problem-oriented teaching model — The traditional problem-oriented teaching model: There will be two PBL case introductions throughout the semester, with face-to-face teaching in physical classrooms.
  Other Names: The control group will accept the traditional problem-oriented teaching model in the professional ethics course, 2 hours /per week, for 18 weeks
  Arms: The traditional problem-oriented teaching model

SUMMARY:
Medical ecology is a highly uncertain and high-pressure environment. Nurses must use their thinking to make critical judgments and decisions in a short time. Since the outbreak of the Covid-19 epidemic, many universities have produced a lot of innovative inf teaching styles. With the reduction of budget and the evaluation of teaching quality, the blended learning model is gradually being valued by educators.

The aims of this study are to establish a teaching model that applies blended learning and problem-oriented teaching, and to explore the association and effectiveness of critical thinking and ethical competence of research subjects after this intervention in which shortens the gap in learning and practicing for increasing clinical nursing capabilities.

DETAILED DESCRIPTION:
Medical ecology is a highly uncertain and high-pressure environment. Nurses must use their thinking to make critical judgments and decisions in a short time. Since the outbreak of the Covid-19 epidemic, many universities have produced a lot of innovative inf teaching styles. With the reduction of budget and the evaluation of teaching quality, the blended learning model is gradually being valued by educators.

The aims of this study are to establish a teaching model that applies blended learning and problem-oriented teaching, and to explore the association and effectiveness of critical thinking and ethical competence of research subjects after this intervention in which shortens the gap in learning and practicing for increasing clinical nursing capabilities.

After the implementation of this protocol, the participants would increase the critical thinking and ethical competence of nursing students in geriatric nursing. Also, the teacher can self-review the teaching effect and analyze the actual situation of the students in the construction of ethical competency as a teaching reference to improve or revise teaching strategies.

ELIGIBILITY:
Inclusion Criteria:

* The research object of this project will be the students in the nursing class of a university (third year students), and the students who have taken 2 credits each of " Profession and Ethics"in two working class.

Exclusion Criteria:

* Students that have selected " Profession and Ethics" but do not wish to participate in this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-01-05 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
The Critical Thinking Disposition Inventory(CTDI-CV) | Baseline (T0)
  This scale is a scale commonly used in education to evaluate critical thinking assessments. There are 18 items in total. The overall internal consistency and retest stability coefficient both exceed 0.8. It has good reliability and validity. The total score ranges from 18 to 108, with higher scores indicating greater critical thinking ability.
Moral distress scale | Baseline (T0)
  This scale is the earliest measurement tool developed in the United States. It can effectively quantify the degree of moral distress generated by nurses when performing care activities. There are 11 questions in total. It can be used to simultaneously measure the frequency of incidents of moral and ethical distress during work and the range of scores. On a scale of 1 (never) to 5 (always), it is also possible to further assess the density of subjects faced with ethically distressing events, with scores ranging from 1 (never) to 5 (many), and when the two are multiplied, which is expressed as the degree of moral and ethical distress. The lower the score, the lower the moral and ethical distress experienced by the nurse in the experience of clinical practice, but the higher the score, the more painful the feelings caused by the moral and ethical distress. higher.
Nurses' Moral Courage Scale，NMCS | Baseline (T0)
  This scale is mainly used to measure the moral courage of clinical nurses' self-assessment. The scale consists of four dimensions and 21 items. They were: ethics (7 items), commitment to good patient care (5 items), compassion and genuine presence with patients (5 items), and ethical responsibility (4 items). Using the Likert 5-point scoring method, "completely disagrees with me" is 1 point, "somewhat disagrees with me" is 2 points, "somewhat agrees with me" is 3 points, "somewhat agrees with me" is 4 points, and "meets me" is 5 points. "Completely agree" is 5 points, and the total scale is 21 to 105 points. The higher the score, the greater the moral courage of the nurse.
The Critical Thinking Disposition Inventory(CTDI-CV) | eighteen weeks after intervention(T1)
  This scale is a scale commonly used in education to evaluate critical thinking assessments. There are 18 items in total. The overall internal consistency and retest stability coefficient both exceed 0.8. It has good reliability and validity. The total score ranges from 18 to 108, with higher scores indicating greater critical thinking ability.
Moral distress scale | eighteen weeks after intervention(T1)
  This scale is the earliest measurement tool developed in the United States. It can effectively quantify the degree of moral distress generated by nurses when performing care activities. There are 11 questions in total. It can be used to simultaneously measure the frequency of incidents of moral and ethical distress during work and the range of scores. On a scale of 1 (never) to 5 (always), it is also possible to further assess the density of subjects faced with ethically distressing events, with scores ranging from 1 (never) to 5 (many), and when the two are multiplied, which is expressed as the degree of moral and ethical distress. The lower the score, the lower the moral and ethical distress experienced by the nurse in the experience of clinical practice, but the higher the score, the more painful the feelings caused by the moral and ethical distress. higher.
Nurses' Moral Courage Scale，NMCS | eighteen weeks after intervention(T1)
  This scale is mainly used to measure the moral courage of clinical nurses' self-assessment. The scale consists of four dimensions and 21 items. They were: ethics (7 items), commitment to good patient care (5 items), compassion and genuine presence with patients (5 items), and ethical responsibility (4 items). Using the Likert 5-point scoring method, "completely disagrees with me" is 1 point, "somewhat disagrees with me" is 2 points, "somewhat agrees with me" is 3 points, "somewhat agrees with me" is 4 points, and "meets me" is 5 points. "Completely agree" is 5 points, and the total scale is 21 to 105 points. The higher the score, the greater the moral courage of the nurse.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Corley MC, Elswick RK, Gorman M, Clor T. Development and evaluation of a moral distress scale. J Adv Nurs. 2001 Jan;33(2):250-6. doi: 10.1046/j.1365-2648.2001.01658.x. PMID 11168709
- [Result] Elrggal ME, Karami NA, Rafea B, Alahmadi L, Al Shehri A, Alamoudi R, Koshak H, Alkahtani S, Cheema E. Evaluation of preparedness of healthcare student volunteers against Middle East respiratory syndrome coronavirus (MERS-CoV) in Makkah, Saudi Arabia: a cross-sectional study. Z Gesundh Wiss. 2018;26(6):607-612. doi: 10.1007/s10389-018-0917-5. Epub 2018 Apr 14. PMID 30533343
- [Result] Han Y, Yang H. The transmission and diagnosis of 2019 novel coronavirus infection disease (COVID-19): A Chinese perspective. J Med Virol. 2020 Jun;92(6):639-644. doi: 10.1002/jmv.25749. Epub 2020 Mar 12. PMID 32141619
- [Result] Hayter M, Jackson D. Pre-registration undergraduate nurses and the COVID-19 pandemic: Students or workers? J Clin Nurs. 2020 Sep;29(17-18):3115-3116. doi: 10.1111/jocn.15317. Epub 2020 May 19. No abstract available. PMID 32369639
- [Result] Hernandez-Martinez A, Rodriguez-Almagro J, Martinez-Arce A, Romero-Blanco C, Garcia-Iglesias JJ, Gomez-Salgado J. Nursing students' experience and training in healthcare aid during the COVID-19 pandemic in Spain. J Clin Nurs. 2021 Feb 15:10.1111/jocn.15706. doi: 10.1111/jocn.15706. Online ahead of print. PMID 33590573
- [Result] Hwang SY, Yen M, Lee BO, Huang MC, Tseng HF. A critical thinking disposition scale for nurses: short form. J Clin Nurs. 2010 Nov;19(21-22):3171-6. doi: 10.1111/j.1365-2702.2010.03343.x. Epub 2010 Sep 8. PMID 21040020
- [Result] Jackson D, Bradbury-Jones C, Baptiste D, Gelling L, Morin K, Neville S, Smith GD. Life in the pandemic: Some reflections on nursing in the context of COVID-19. J Clin Nurs. 2020 Jul;29(13-14):2041-2043. doi: 10.1111/jocn.15257. Epub 2020 Apr 12. No abstract available. PMID 32281185
- [Result] Khodaveisi M, Oshvandi K, Bashirian S, Khazaei S, Gillespie M, Masoumi SZ, Mohammadi F. Moral courage, moral sensitivity and safe nursing care in nurses caring of patients with COVID-19. Nurs Open. 2021 Nov;8(6):3538-3546. doi: 10.1002/nop2.903. Epub 2021 May 4. PMID 33945661
- [Result] Liu Y, Yan LM, Wan L, Xiang TX, Le A, Liu JM, Peiris M, Poon LLM, Zhang W. Viral dynamics in mild and severe cases of COVID-19. Lancet Infect Dis. 2020 Jun;20(6):656-657. doi: 10.1016/S1473-3099(20)30232-2. Epub 2020 Mar 19. No abstract available. PMID 32199493
- [Result] Robertson DW. Ethical theory, ethnography, and differences between doctors and nurses in approaches to patient care. J Med Ethics. 1996 Oct;22(5):292-9. doi: 10.1136/jme.22.5.292. PMID 8910782
- [Result] Strang P, Martinsson L, Bergstrom J, Lundstrom S. COVID-19: Symptoms in Dying Residents of Nursing Homes and in Those Admitted to Hospitals. J Palliat Med. 2021 Jul;24(7):1067-1071. doi: 10.1089/jpm.2020.0688. Epub 2021 Mar 5. PMID 33667124
- [Result] Swift A, Banks L, Baleswaran A, Cooke N, Little C, McGrath L, Meechan-Rogers R, Neve A, Rees H, Tomlinson A, Williams G. COVID-19 and student nurses: A view from England. J Clin Nurs. 2020 Sep;29(17-18):3111-3114. doi: 10.1111/jocn.15298. Epub 2020 May 15. No abstract available. PMID 32298512
- [Result] Tuijt R, Frost R, Wilcock J, Robinson L, Manthorpe J, Rait G, Walters K. Life under lockdown and social restrictions - the experiences of people living with dementia and their carers during the COVID-19 pandemic in England. BMC Geriatr. 2021 May 10;21(1):301. doi: 10.1186/s12877-021-02257-z. PMID 33971847
- [Result] van der Dam S, Abma TA, Kardol MJ, Widdershoven GA. "Here's my dilemma". Moral case deliberation as a platform for discussing everyday ethics in elderly care. Health Care Anal. 2012 Sep;20(3):250-67. doi: 10.1007/s10728-011-0185-9. PMID 21809142
- [Result] Whitehead BR, Torossian E. Older Adults' Experience of the COVID-19 Pandemic: A Mixed-Methods Analysis of Stresses and Joys. Gerontologist. 2021 Jan 21;61(1):36-47. doi: 10.1093/geront/gnaa126. PMID 32886764
- [Result] Yeung DY, Chung EKH, Lam AHK, Ho AKK. Effects of subjective successful aging on emotional and coping responses to the COVID-19 pandemic. BMC Geriatr. 2021 Feb 17;21(1):128. doi: 10.1186/s12877-021-02076-2. PMID 33596829
- [Result] Zou L, Ruan F, Huang M, Liang L, Huang H, Hong Z, Yu J, Kang M, Song Y, Xia J, Guo Q, Song T, He J, Yen HL, Peiris M, Wu J. SARS-CoV-2 Viral Load in Upper Respiratory Specimens of Infected Patients. N Engl J Med. 2020 Mar 19;382(12):1177-1179. doi: 10.1056/NEJMc2001737. Epub 2020 Feb 19. No abstract available. PMID 32074444
- See also: 6 blended learning models: When blended learning is what's up for successful students. — http://elearningindustry.com/6-blended-learning-models-blended-learning-successful-students